CLINICAL TRIAL: NCT02681016
Title: Prospective rAndomized, Single-blind, multicenTral Control Clinical Trial of Sirolimus-eluting coRonary Stent "Calypso" (Angioline) vs Everolimus-elutIng cOronary stenT "Xience Prime" (Abbott Vascular)
Brief Title: Sirolimus-eluting Stent CALYPSO vs Everolimus-eluting Stent XIENCE
Acronym: PATRIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAT1.0
Record Dates: First submitted 2016-01-19; First posted 2016-02-12 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Ischemic Heart Disease; Coronary Atherosclerosis; Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Calypso; Xience; Coronary stenosis; Drug-eluting stent; Coronary angioplasty with stenting; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Coronary Stenosis | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus-eluting stent "Calypso" (Experimental): Commercially approved coronary stent system "Calypso" (Angioline, Russia) Coating - Sirolimus(rapamicine) Stent diameters: 2.0, 2.25, 2.5, 2.75, 3.0, 3.5, 4.0, 4.5 mm. Stent lengths: 8, 13, 15, 18, 23, 28, 33, 38 mm.
  Interventions: Device: DES "Calypso"; Procedure: Coronary angioplasty
- Everolimus-eluting stent "Xience Prime" (Active Comparator): Commercially approved XIENCE PRIME, (Abbott Vascular, USA) Coating - Everolimus with concentration Stent diameters: 2.25, 2.5, 2.75, 3.0, 3.5, 4.0 mm. Stent lengths: 8, 12, 15, 18, 23, 28, 33, 38 mm.
  Interventions: Device: DES "Xience Prime"; Procedure: Coronary angioplasty

INTERVENTIONS:
Device: DES "Calypso" — A standard endovascular procedure is carried out under local anesthesia and under fluoroscopic control. Stenosis of coronary artery is passed by the hydrophilic coronary wire. Then balloon angioplasty of target lesion (if required) is provided. After the angiographic control coronary stent is implanted. After coronary wire removing control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix(clopidogrel) in dose 300-600 mg prescription before the procedure and heparin (heparin sodium) injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix(clopidogrel) in dose 75/d should be prescribed within 12 months.
  Arms: Sirolimus-eluting stent "Calypso"
Device: DES "Xience Prime" — A standard endovascular procedure is carried out under local anesthesia and under fluoroscopic control. Stenosis of coronary artery is passed by the hydrophilic coronary wire. Then balloon angioplasty of target lesion (if required) is provided. After the angiographic control coronary stent is implanted. After coronary wire removing control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix(clopidogrel) in dose 300-600 mg prescription before the procedure and heparin (heparin sodium) injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix(clopidogrel) in dose 75/d should be prescribed within 12 months.
  Arms: Everolimus-eluting stent "Xience Prime"
Procedure: Coronary angioplasty

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of sirolimus-eluting coronary stent "Calypso" (Angioline, Russia) in comparison with everolimus-eluting coronary stent "Xience" (Abbott Vascular, USA)

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for coronary angioplasty with stenting due to Ischemic heart disease (Stable angina, Unstable angina, non-ST Myocardial Infarction).
* Target vessel lesion in coronary artery with diameter measurements >2.5 mm & < 4.5 mm.
* Signed, documented informed consent prior to admission to the study

Exclusion Criteria:

* Age <18 years or >75 years
* Renal insufficiency (GFR/MDRD <30 ml/min)
* Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
* Known non-adherence to DAPT
* LVEF <30%
* Known oncology
* Severe cardiac valvular pathology, requiring operative treatment within 1 year
* Anemia (HB<100 g/l)
* Continuing bleeding
* Acute coronary syndrome (ST-elevation Myocardial infarction)
* Anamnesis of previous coronary angioplasty/stenting or CABG
* NYHA class (dyspnoea) IV or hospitalization during last year due to Chronic cardiac failure as a primary diagnosis.
* Pregnancy
* Coronary pathology requiring CABG or staged scheduled coronary angioplasty/stenting except cases of unscheduled staged coronary angioplasty/stenting within 4 weeks after primary procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | during 1 year after procedure
  Primary outcome is defined as a composite endpoint of cardiac death, target vessel myocardial infarction and clinically indicated target lesion revascularization.

SECONDARY OUTCOMES:
1 year major adverse cardiac and cerebrovascular events (MACCE) | during 1 year after procedure
  1 year major adverse cardiac and cerebrovascular events (MACCE) including: All-cause mortality, Myocardial infarction, Stroke, Stent thrombosis, Clinically indicated Target lesion revascularization, Any target lesion revascularization, Any target vessel revascularization.

OTHER OUTCOMES:
Angiographic endpoint | 1 year after procedure
  Estimation of target lesion late lumen loss in randomly selected 20% of the subjects.
Device success | procedure
  Device success is defined as achievement of a final residual diameter stenosis 20% during the initial procedure.
Lesion success | procedure
  Lesion success, defined as achievement of a final residual diameter stenosis 20% with use of any PCI approach.
In-hospital procedure success | Within 5-day hospitalization
  Procedure success is defined as achievement of a final residual diameter stenosis 20% together with the absence of any in-hospital major adverse cardiac event. The 5-day hospitalization time frame was evaluated according to the standards of health care in patients was coronary angioplasty in Russia.

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided